CLINICAL TRIAL: NCT04732611
Title: Effects of Pilates Exercises Versus Walking on Mechanical and Vascular Variables of Individuals With Type 2 Diabetes Mellitus: Randomized Clinical Trial
Brief Title: Effects of Pilates Exercises Versus Walking on Mechanical and Vascular Variables of Individuals With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jefferson Fagundes Loss, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 39137
Record Dates: First submitted 2021-01-17; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pilates; Walking; Neuromuscular Adaptation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): Pilates group participants will perform 3 weekly Pilates sessions lasting approximately 50 minutes for 20 weeks.
  Interventions: Other: Pilates exercises
- Walking (Active Comparator): Walking group participants will perform 3 weekly walking sessions lasting approximately 50 minutes for 20 weeks
  Interventions: Other: Walking protocol

INTERVENTIONS:
Other: Pilates exercises — Pilates group participants will perform 3 weekly Pilates sessions lasting approximately 50 minutes for 20 weeks.
  Arms: Pilates
Other: Walking protocol — Walking group participants will perform 3 weekly walking sessions lasting approximately 50 minutes for 20 weeks.
  Arms: Walking

SUMMARY:
The Diabetes Mellitus (DM) is a major worldwide public health problem. The hyperglycemia resulting from DM could lead to metabolic adaptations and physiological changes in different body systems. The DM patients are usually sedentary, once the symptoms as the sensory deficits compromise balance and gait. Giving that this sedentary lifestyle needs to be reversed, since physical exercise is well known a fundamental element in the treatment and prevention of the DM.

The major recommendations to this population is the practice of aerobic exercises and the strength training focused on the biggest muscle groups. It is well know that this type of exercise can improve the uptake of intramuscular glucose. In that context the Pilates Method seems as a good option of exercise, once the method works in a global way, working on different muscle groups in the same exercise. Besides that, to the best of our knowledge there aren't enough studies to support the Pilates Method as an alternative type exercise to help in the glycemic control and in the management of this kind of patients. The aim of this study is to evaluate the efficacy and safety of an exercise program using the Pilates Method versus a walking program in neuromuscular, metabolic and vascular variables in type 2 diabetic patients.

60 participants will be recruited by convenience. Individuals will be eligible if [1] they had type 2 diabetes mellitus; [2] men and women aged 35 to 60 years [3] medical approval to practice exercise; [4] do not have any bone, joint or muscle disease that make the practice of exercises impossible; [5] not being pregnant; [6] not being unable to follow the instructions for any reason and [7] at least 6 months without exercising. The participants' eligibility will be checked by the researcher. Subsequently, they will be allocated randomly in one of the two groups (Pilates Group or Walking).

Pilates group participants will perform 3 Pilates sessions a week lasting approximately 50 minutes for 20 weeks. Walking group participants will perform 3 walking sessions a week lasting approximately 50 minutes for 20 weeks. All the exercises sessions will be supervised by a professional.

All the participants will be evaluated at the baseline and after 20 weeks of exercises. The main outcome of this study are the Triceps surae muscle force and the blood glycose. The secondary outcomes are Triceps surae muscle architecture, mechanical adaptations of the Achilles tendon and endothelial function.

Our hypothesis is that both groups will be safety and efficiency to improve the Triceps surae muscle force and to decrease blood glycose. Our secondary hypothesis is that the Pilates Group will show better results to both primary outcomes than the walking group.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Men and women between 35 and 65 years old;
* Possess type 2 diabetes mellitus diagnosed;
* Medical approval to practice exercise;
* Do not have any bone, joint or muscle disease that make impossible do the exercises;
* not being pregnant;
* not being unable to follow the instructions for any reason;
* not be exercising for at least 6 months.

Exclusion Criteria:

* Incapacity to follow the instructions for any reason;
* Beginning another treatment for DM2, either physical therapy, exercises or changes of the medical care throughout the study period.
* Having practiced exercises in the last six months;
* Pregnancy;

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Triceps surae muscle force | 20 weeks
  Triceps surae muscle force assessed by isokinetic dynamometry.
Blood Glycose | 20 weeks
  Blood Glycose assessed by HbA1c

SECONDARY OUTCOMES:
Triceps surae muscle architecture | 20 weeks
  Triceps surae muscle architecture assessed by ultrasound
Mechanical adaptations of the Achilles tendon | 20 weeks
  Mechanical adaptations of the Achilles tendon assessed by ultrasound
Endothelial function | 20 weeks
  Endothelial function assessed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson F Loss, PhD, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akashi PM, Sacco IC, Watari R, Hennig E. The effect of diabetic neuropathy and previous foot ulceration in EMG and ground reaction forces during gait. Clin Biomech (Bristol). 2008 Jun;23(5):584-92. doi: 10.1016/j.clinbiomech.2007.11.015. Epub 2008 Feb 21. PMID 18178296
- [Background] American College of Sports Medicine. Diretrizes do ACSM para os testes de esforço e sua prescrição. 9 ed. - Rio de Janeiro: Guanabara, 2017
- [Background] Andersen H, Nielsen S, Mogensen CE, Jakobsen J. Muscle strength in type 2 diabetes. Diabetes. 2004 Jun;53(6):1543-8. doi: 10.2337/diabetes.53.6.1543. PMID 15161759
- [Background] Arya S, Kulig K. Tendinopathy alters mechanical and material properties of the Achilles tendon. J Appl Physiol (1985). 2010 Mar;108(3):670-5. doi: 10.1152/japplphysiol.00259.2009. Epub 2009 Nov 5. PMID 19892931
- [Background] Bacarin TA, Sacco IC, Hennig EM. Plantar pressure distribution patterns during gait in diabetic neuropathy patients with a history of foot ulcers. Clinics (Sao Paulo). 2009;64(2):113-20. doi: 10.1590/s1807-59322009000200008. PMID 19219316
- [Background] Baroni BM, Geremia JM, Rodrigues R, De Azevedo Franke R, Karamanidis K, Vaz MA. Muscle architecture adaptations to knee extensor eccentric training: rectus femoris vs. vastus lateralis. Muscle Nerve. 2013 Oct;48(4):498-506. doi: 10.1002/mus.23785. Epub 2013 Jul 15. PMID 23852989
- [Background] Batista F, Nery C, Pinzur M, Monteiro AC, de Souza EF, Felippe FH, Alcantara MC, Campos RS. Achilles tendinopathy in diabetes mellitus. Foot Ankle Int. 2008 May;29(5):498-501. doi: 10.3113/FAI-2008-0498. PMID 18510903
- [Background] Bayat F, Shojaeezadeh D, Baikpour M, Heshmat R, Baikpour M, Hosseini M. The effects of education based on extended health belief model in type 2 diabetic patients: a randomized controlled trial. J Diabetes Metab Disord. 2013 Oct 28;12(1):45. doi: 10.1186/2251-6581-12-45. PMID 24517170
- [Background] Bland's, M. (2009).
- [Background] Blazevich AJ. Effects of physical training and detraining, immobilisation, growth and aging on human fascicle geometry. Sports Med. 2006;36(12):1003-17. doi: 10.2165/00007256-200636120-00002. PMID 17123325
- [Background] Caselli A, Pham H, Giurini JM, Armstrong DG, Veves A. The forefoot-to-rearfoot plantar pressure ratio is increased in severe diabetic neuropathy and can predict foot ulceration. Diabetes Care. 2002 Jun;25(6):1066-71. doi: 10.2337/diacare.25.6.1066. PMID 12032116
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement executive summary. Diabetes Care. 2010 Dec;33(12):2692-6. doi: 10.2337/dc10-1548. No abstract available. PMID 21115771
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] SILVA, N. R.; COSTA, C. E. M. A hiperglicemia e os mecanismos envolvidos nas disfunções vasculares do Diabetes Mellitus. Arq. Ciênc.Saúde Unipar, Umuarama, v. 12, n. 3, p. 265-270, set./dez. 2008
- [Background] Dekerle J, Baron B, Dupont L, Vanvelcenaher J, Pelayo P. Maximal lactate steady state, respiratory compensation threshold and critical power. Eur J Appl Physiol. 2003 May;89(3-4):281-8. doi: 10.1007/s00421-002-0786-y. Epub 2003 Mar 4. PMID 12736836
- [Background] DIABETES CARE. American Diabetes Association. Diagnosis and classification of diabetes mellitus. 2014.
- [Background] Esformes JI, Narici MV, Maganaris CN. Measurement of human muscle volume using ultrasonography. Eur J Appl Physiol. 2002 May;87(1):90-2. doi: 10.1007/s00421-002-0592-6. Epub 2002 Mar 27. PMID 12012082
- [Background] Fang M. Trends in Diabetes Management Among US Adults: 1999-2016. J Gen Intern Med. 2020 May;35(5):1427-1434. doi: 10.1007/s11606-019-05587-2. Epub 2020 Jan 2. PMID 31898135
- [Background] Farinha JB, Ramis TR, Vieira AF, Macedo RCO, Rodrigues-Krause J, Boeno FP, Schroeder HT, Muller CH, Boff W, Krause M, De Bittencourt PIH Jr, Reischak-Oliveira A. Glycemic, inflammatory and oxidative stress responses to different high-intensity training protocols in type 1 diabetes: A randomized clinical trial. J Diabetes Complications. 2018 Dec;32(12):1124-1132. doi: 10.1016/j.jdiacomp.2018.09.008. Epub 2018 Sep 19. PMID 30270019
- [Background] Ferguson B. ACSM's Guidelines for Exercise Testing and Prescription 9th Ed. 2014. J Can Chiropr Assoc. 2014 Sep;58(3):328.
- [Background] Fernando ME, Crowther RG, Lazzarini PA, Sangla KS, Wearing S, Buttner P, Golledge J. Plantar pressures are higher in cases with diabetic foot ulcers compared to controls despite a longer stance phase duration. BMC Endocr Disord. 2016 Sep 15;16(1):51. doi: 10.1186/s12902-016-0131-9. PMID 27629263
- [Background] Ferreira MC, Tozatti J, Fachin SM, Oliveira PP, Santos RF, Silva ME. [Reduction of functional mobility and cognitive capacity in type 2 diabetes mellitus]. Arq Bras Endocrinol Metabol. 2014 Dec;58(9):946-52. doi: 10.1590/0004-2730000003097. Portuguese. PMID 25627051
- [Background] Fowler MJ. Microvascular and macrovascular complications of diabetes. Clin Diabetes. 2008;26(2):77-82
- [Background] Geremia JM, Bobbert MF, Casa Nova M, Ott RD, Lemos Fde A, Lupion Rde O, Frasson VB, Vaz MA. The structural and mechanical properties of the Achilles tendon 2 years after surgical repair. Clin Biomech (Bristol). 2015 Jun;30(5):485-92. doi: 10.1016/j.clinbiomech.2015.03.005. Epub 2015 Mar 11. PMID 25828432
- [Background] Giacomozzi C, Sartor CD, Telles R, Uccioli L, Sacco ICN. Ulcer-risk classification and plantar pressure distribution in patients with diabetic polyneuropathy: exploring the factors that can lead to foot ulceration. Ann Ist Super Sanita. 2018 Oct-Dec;54(4):284-293. doi: 10.4415/ANN_18_04_04. PMID 30575564
- [Background] Gomes AA, Onodera AN, Otuzi ME, Pripas D, Mezzarane RA, Sacco IC. Electromyography and kinematic changes of gait cycle at different cadences in diabetic neuropathic individuals. Muscle Nerve. 2011 Aug;44(2):258-68. doi: 10.1002/mus.22051. PMID 21755508
- [Background] Kawakami Y, Abe T, Fukunaga T. Muscle-fiber pennation angles are greater in hypertrophied than in normal muscles. J Appl Physiol (1985). 1993 Jun;74(6):2740-4. doi: 10.1152/jappl.1993.74.6.2740. PMID 8365975
- [Background] Lemaster JW, Reiber GE, Smith DG, Heagerty PJ, Wallace C. Daily weight-bearing activity does not increase the risk of diabetic foot ulcers. Med Sci Sports Exerc. 2003 Jul;35(7):1093-9. doi: 10.1249/01.MSS.0000074459.41029.75. PMID 12840628
- [Background] Mademli L, Arampatzis A. Behaviour of the human gastrocnemius muscle architecture during submaximal isometric fatigue. Eur J Appl Physiol. 2005 Aug;94(5-6):611-7. doi: 10.1007/s00421-005-1366-8. Epub 2005 May 20. PMID 15906075
- [Background] Magnusson SP, Aagaard P, Dyhre-Poulsen P, Kjaer M. Load-displacement properties of the human triceps surae aponeurosis in vivo. J Physiol. 2001 Feb 15;531(Pt 1):277-88. doi: 10.1111/j.1469-7793.2001.0277j.x. PMID 11179410
- [Background] Martinelli AR, Mantovani AM, Nozabieli AJ, Ferreira DM, Barela JA, Camargo MR, Fregonesi CE. Muscle strength and ankle mobility for the gait parameters in diabetic neuropathies. Foot (Edinb). 2013 Mar;23(1):17-21. doi: 10.1016/j.foot.2012.11.001. Epub 2012 Dec 27. PMID 23274122
- [Background] Musi N, Fujii N, Hirshman MF, Ekberg I, Froberg S, Ljungqvist O, Thorell A, Goodyear LJ. AMP-activated protein kinase (AMPK) is activated in muscle of subjects with type 2 diabetes during exercise. Diabetes. 2001 May;50(5):921-7. doi: 10.2337/diabetes.50.5.921. PMID 11334434
- [Background] Narici M. Human skeletal muscle architecture studied in vivo by non-invasive imaging techniques: functional significance and applications. J Electromyogr Kinesiol. 1999 Apr;9(2):97-103. doi: 10.1016/s1050-6411(98)00041-8. PMID 10098710
- [Background] OLIVEIERA, S. G.; ZUGNO, R.; SILVA, P. C. The incidence of type 1 diabetes mellitus in southern Brazil. Revista Saúde e Desenvolvimento, v.13, n.15, 2019.
- [Background] OLIVEIRA, J. E. P.; VENCIO, S. Diretrizes da Sociedade Brasileira de Diabetes: 2014-2015/ Sociedade Brasileira de Diabetes, São Paulo: AC Farmacêutica, 2015.
- [Background] Parastesh M, Heidarianpour A, Sadegh M. Investigating the effects of endurance, resistance and combined training on reproductive hormones and sperm parameters of streptozotocin-nicotinamide diabetic male rats. J Diabetes Metab Disord. 2019 Jun 19;18(2):273-279. doi: 10.1007/s40200-018-0380-4. eCollection 2019 Dec. PMID 31890651
- [Background] Pasnoor M, Dimachkie MM, Kluding P, Barohn RJ. Diabetic neuropathy part 1: overview and symmetric phenotypes. Neurol Clin. 2013 May;31(2):425-45. doi: 10.1016/j.ncl.2013.02.004. Epub 2013 Mar 15. PMID 23642717
- [Background] Picon AP, Ortega NR, Watari R, Sartor C, Sacco IC. Classification of the severity of diabetic neuropathy: a new approach taking uncertainties into account using fuzzy logic. Clinics (Sao Paulo). 2012;67(2):151-6. doi: 10.6061/clinics/2012(02)10. PMID 22358240
- [Background] Qiu S, Cai X, Schumann U, Velders M, Sun Z, Steinacker JM. Impact of walking on glycemic control and other cardiovascular risk factors in type 2 diabetes: a meta-analysis. PLoS One. 2014 Oct 17;9(10):e109767. doi: 10.1371/journal.pone.0109767. eCollection 2014. PMID 25329391
- [Background] Richardson JK. Factors associated with falls in older patients with diffuse polyneuropathy. J Am Geriatr Soc. 2002 Nov;50(11):1767-73. doi: 10.1046/j.1532-5415.2002.50503.x. PMID 12410893
- [Background] Sacco IC, Hamamoto AN, Onodera AN, Gomes AA, Weiderpass HA, Pachi CG, Yamamoto JF, von Tscharner V. Motor strategy patterns study of diabetic neuropathic individuals while walking. A wavelet approach. J Biomech. 2014 Jul 18;47(10):2475-82. doi: 10.1016/j.jbiomech.2014.04.007. Epub 2014 Apr 19. PMID 24816334
- [Background] SACCO ICN, SARTOR CD, GOMES AA, JOÃO SMA, E CRONFLI R. Avaliação das perdas sensório-motoras do pé e tornozelo decorrentes da neuropatia diabética. Rev. Bras. Fisioter., São Carlos, v. 11, n. 1, p. 27-33, jan./fev. 2007
- [Background] Sacco IC, Akashi PM, Hennig EM. A comparison of lower limb EMG and ground reaction forces between barefoot and shod gait in participants with diabetic neuropathic and healthy controls. BMC Musculoskelet Disord. 2010 Feb 3;11:24. doi: 10.1186/1471-2474-11-24. PMID 20128894
- [Background] Salsich GB, Brown M, Mueller MJ. Relationships between plantar flexor muscle stiffness, strength, and range of motion in subjects with diabetes-peripheral neuropathy compared to age-matched controls. J Orthop Sports Phys Ther. 2000 Aug;30(8):473-83. doi: 10.2519/jospt.2000.30.8.473. PMID 10949504
- [Background] Sawacha Z, Spolaor F, Guarneri G, Contessa P, Carraro E, Venturin A, Avogaro A, Cobelli C. Abnormal muscle activation during gait in diabetes patients with and without neuropathy. Gait Posture. 2012 Jan;35(1):101-5. doi: 10.1016/j.gaitpost.2011.08.016. Epub 2011 Nov 17. PMID 22098824
- [Background] Schalkwijk CG, Stehouwer CD. Vascular complications in diabetes mellitus: the role of endothelial dysfunction. Clin Sci (Lond). 2005 Aug;109(2):143-59. doi: 10.1042/CS20050025. PMID 16033329
- [Background] Scheffel RS, Bortolanza D, Weber CS, Costa LA, Canani LH, Santos KG, Crispim D, Roisenberg I, Lisboa HR, Tres GS, Tschiedel B, Gross JL. [Prevalence of micro and macroangiopatic chronic complications and their risk factors in the care of out patients with type 2 diabetes mellitus]. Rev Assoc Med Bras (1992). 2004 Jul-Sep;50(3):263-7. doi: 10.1590/s0104-42302004000300031. Epub 2004 Oct 21. Portuguese. PMID 15499476
- [Background] Schmidt MI, Hoffmann JF, de Fatima Sander Diniz M, Lotufo PA, Griep RH, Bensenor IM, Mill JG, Barreto SM, Aquino EM, Duncan BB. High prevalence of diabetes and intermediate hyperglycemia - The Brazilian Longitudinal Study of Adult Health (ELSA-Brasil). Diabetol Metab Syndr. 2014 Nov 18;6:123. doi: 10.1186/1758-5996-6-123. eCollection 2014. PMID 25788987
- [Background] SENIAM. (2017). Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles. Retrieved from http://www.seniam.org/
- [Background] Sinacore DR, Gutekunst DJ, Hastings MK, Strube MJ, Bohnert KL, Prior FW, Johnson JE. Neuropathic midfoot deformity: associations with ankle and subtalar joint motion. J Foot Ankle Res. 2013 Mar 25;6(1):11. doi: 10.1186/1757-1146-6-11. PMID 23531372
- [Background] SOCIEDADE BRASILEIRA DE DIABETES. Diretrizes Sociedade Brasileira de Diabetes 2017-2018, p.19-26, 2018.
- [Background] Souza C, Kruger RL, Schmit EFD, Wagner Neto ES, Reischak-Oliveira A, de Sa CKC, Loss JF. Cardiorespiratory Adaptation to Pilates Training. Res Q Exerc Sport. 2021 Sep;92(3):453-459. doi: 10.1080/02701367.2020.1749222. Epub 2020 Jun 4. PMID 32493165
- [Background] Suda EY, Madeleine P, Hirata RP, Samani A, Kawamura TT, Sacco IC. Reduced complexity of force and muscle activity during low level isometric contractions of the ankle in diabetic individuals. Clin Biomech (Bristol). 2017 Feb;42:38-46. doi: 10.1016/j.clinbiomech.2017.01.001. Epub 2017 Jan 4. PMID 28088014
- [Background] Thurman DJ, Stevens JA, Rao JK; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: Assessing patients in a neurology practice for risk of falls (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2008 Feb 5;70(6):473-9. doi: 10.1212/01.wnl.0000299085.18976.20. PMID 18250292
- [Background] Veves A, Murray HJ, Young MJ, Boulton AJ. The risk of foot ulceration in diabetic patients with high foot pressure: a prospective study. Diabetologia. 1992 Jul;35(7):660-3. doi: 10.1007/BF00400259. PMID 1644245
- [Background] Watari R, Sartor CD, Picon AP, Butugan MK, Amorim CF, Ortega NR, Sacco IC. Effect of diabetic neuropathy severity classified by a fuzzy model in muscle dynamics during gait. J Neuroeng Rehabil. 2014 Feb 8;11:11. doi: 10.1186/1743-0003-11-11. PMID 24507153